CLINICAL TRIAL: NCT04927871
Title: Hybridized Three Steps (HITS) Intervention to Prevent Diabetes in Venezuela: HITS Diabetes With Prevention, An EVESCAM Lifestyle Intervention Study
Brief Title: Hybridized Three Steps Intervention to Prevent Diabetes in Venezuela
Acronym: HITS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation for Public Health and Epidemiological Research of Venezuela (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FISPEVEN
Record Dates: First submitted 2021-02-15; First posted 2021-06-16 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Obesity; Overweight; PreDiabetes; Diabetes Mellitus, Type 2; Risk Factor, Cardiovascular
MeSH Terms: conditions — Obesity; Overweight; Prediabetic State; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hybridized Lyfestile Intervention (Experimental): The participants will receive three interventions including Total Diet Replacement, Medical Nutrition Therapy, and the Diabetes Prevention Program
  Interventions: Behavioral: Total Diet Replacement (TDR); Behavioral: Medical Nutritional Therapy (MNT); Behavioral: Diabetes Prevention Program 4 months
- Only Diabetes Prevention Program (Active Comparator): The comparison group will receive only the Diabetes Prevention Program
  Interventions: Behavioral: Diabetes Prevention Program

INTERVENTIONS:
Behavioral: Total Diet Replacement (TDR) — The nutritionist will provide a total diet replacement (TDR) with Low-Energy Liquid-Diet (LELD - 811 kcal/day, 64 g protein, 132 g carbohydrate, 6 g fat) and the food reintroduction for two months.
  Arms: Hybridized Lyfestile Intervention
Behavioral: Medical Nutritional Therapy (MNT) — The nutritionist will provide Medical Nutritional Therapy (MNT) using the transcultural Diabetes Nutritional Algorithm (tDNA) Toolkit adapted for Venezuela for four months.
  Arms: Hybridized Lyfestile Intervention
Behavioral: Diabetes Prevention Program 4 months — The coach will provide a group-based Diabetes Prevention Program (DPP) version in weekly encounters during 4-months.
  Arms: Hybridized Lyfestile Intervention
Behavioral: Diabetes Prevention Program — The coach will provide a group-based Diabetes Prevention Program (DPP) version in weekly encounters during 6-months.
  Arms: Only Diabetes Prevention Program

SUMMARY:
The American Diabetes Association recommends implementing the Diabetes Prevention Program (DPP) in subjects with prediabetes. In the DPP, weight reduction was the main predictor of a lower incidence of type 2 diabetes (T2D), each kilogram lost was related with 16% lower incidence. However, the effectiveness of the DPP in primary care settings is lower than the original study. A meta-analysis of 36 pragmatic clinical trials of DPP in primary care settings showed a reduction in T2D incidence by 26%, less than half than the original study (58%), with a pooled mean weight loss 1.57 kg higher than standard care, demonstrating the large difficulties to reduce weight of participants at community levels. Total diet replacement (TDR) with low-energy liquid-diet or solid diet (825-853 kcal/day) is an effective strategy to reduce weight. The effectiveness of an intervention including initial rapid weight loss before starting the DPP is ignored in primary care levels in Venezuela. We aim: 1- To compare the weight loss achieved of two lifestyle intervention programs in a community health center of Venezuela: a) A hybrid lifestyle including rapid weight loss with total diet replacement (TDR), then medical nutrition therapy (MNT), and the DPP, VS b) only the DPP; 2- To evaluate the change of cardiometabolic risk factors between groups; 3- To evaluate the implementation process. Our hypothesis is: after six months of intervention, subjects receiving a hybridized lifestyle (TDR+MNT+DPP) will double the weight loss of those that only receive DPP.

DETAILED DESCRIPTION:
In Venezuela, mortality for cardiovascular disease (CVD) was responsible for 30.5% of all deaths, increasing by 8.3% since 2007 to 2017. The prevalence of cardiometabolic risk factors in the country is also increasing. The investigators led two cross-sectional surveys in Venezuela, the VEMSOLS, evaluating 1320 adults between 2006 to 2010, and the EVESCAM, a national representative sample of 3420 adults, from 2014 to 20178, and the change of cardiometabolic risk factors prevalence was hypertension from 30.0% to 34.1%, metabolic syndrome from 35.7% to 42.2%, diabetes from 8.0% to 12.3%, and prediabetes from 14.4% to 34.9%. Prediabetes increased 242% in a decade, from 2.4 to 7 million of adults, estimating that 1.7 million of adults could advance to type 2 diabetes (T2D) in the next 3 to 5 years The American Diabetes Association recommends implementing the Diabetes Prevention Program (DPP) in subjects with prediabetes. This program aims weight reduction increasing physical activity and healthy eating. In controlled settings, DPP has consistently proved to reduce T2D incidence by 58%, with long term benefits. However, to translate this effectiveness to primary care settings is a major challenge. In Latin America, two studies on T2D prevention were done at the same time, funded by an International Diabetes Federation (IDF) initiative, with contradictory results. In Venezuela, Florez et al. implemented a Randomized Controlled Trial (RCT) using the US-DPP version, with a multidisciplinary team, on 140 adults with prediabetes and overweight, to receive standard care vs. lifestyle intervention (LSI), during two-years. LSI group lost more than 10% of basal weight compared with 2.3% in the standard care group (p< 0.001), none developed T2D compared with 6% of the crude cumulative incidence of T2D in the standard care group (p<0.05)15, and lipid profile and cardiovascular health score also improved. Contrarily, in Colombia, Barengo et al implemented the Finnish Diabetes Prevention Study (DPS) in primary health care centers, provided by specialists in physical activity and nutritionists on 772 adults with prediabetes, randomly assigned to LSI vs. standard care during two-years. Metabolic components, reversion to normoglycemia and T2D incidence were similar between groups. A meta-analysis of 36 pragmatic clinical trials of diabetes prevention programs in primary care settings showed a reduction in T2D incidence by 26%, less than half than the original studies (58%). In these studies LSI only showed a pooled mean weight loss 1.57 kg higher than standard care, demonstrating the large difficulties to reduce the weight of participants at community levels.

The team is leading in Venezuela a transculturalization process incorporating multiple validated components to significantly improve the effectiveness of preventive medicine initiatives for T2D, and by extension, positively impact T2D incidence, prevalence, quality of life, and health care costs.

To prevent T2D effectively, LSI programs need to induce weight loss. In the DPP, weight reduction was the main predictor of a lower incidence of T2D, each kilogram lost was related with 16% lower incidence. Total diet replacement (TDR) with low-energy liquid-diet or solid diet (825-853 kcal/day) is an effective strategy to reduce weight. In the PREVIEW study, 2224 participants with prediabetes and obesity received a low energy diet during 8-week and presented a mean weight loss of 10.7 ± 0.4 kg, and 83.5% achieved the target of ≥8% weight reduction, and expected incidence of T2D at three-year was only 4%, independent on the intervention used post-weight-loss. However, the effectiveness of intervention including an initial rapid weight loss in primary care levels in Venezuela is ignored. In order to improve the effectiveness of T2D prevention programs the following objectives are proposed:

1. To compare the weight loss achieved with two LSI programs in a community health center of Venezuela: a) A hybrid LSI including rapid weight loss with total diet replacement (TDR), followed by medical nutrition therapy (MNT), and the DPP protocol, vs b) only the DPP.
2. To compare the change of cardiometabolic risk factors between groups.
3. To evaluate the implementation process.

The hypothesis is: after six months of intervention, subjects receiving a hybridized LSI (TDR+MNT+DPP) will double the weight loss of those that only receive DPP (This is based on the pilot study - see below). If this outcome is achieved, it will have an enormous impact in the way that the DPP should be provided in the primary health care systems in developing countries, increasing the effectiveness of weight reduction, and in consequence, improving cardiovascular health.

Approach Design: A pragmatic mix trial was designed with two groups a) subjects receiving a hybridized LSI (TDR-MNT-DPP) and b) only DPP.

Sampling: Community members will be invited to a medical screening at the community health care center. Those with high risk will be identified using the Latin America Finish Diabetes Risk Score (LA-FINRISC). The LA-FINDRISC is a non-invasive tool that includes age, body mass index (BMI), waist circumference, physical activity, daily consumption of fruits and vegetables, history of hyperglycemia, history of antihypertensive drug treatment, and family history of diabetes, assigning a score ranging from 0 to 26 points. In Venezuelan adults, 9 points are the best score (sensitivity 71.4% + specificity 65.4%) to detect subjects with impaired glucose tolerance. Those with an LA-FINDRISC ≥ 10 points and having the inclusion criteria will be invited to laboratory test and medical evaluation and those with laboratory criteria will be invited to participate.

Sample Size: The formula to compare two mean was used. Based on preliminary results of the pilot study, the aim was to detect a two-fold reduction of weight loss in the intensive group (mean = 5.0 kg, standard deviation = 4.9) compared with only DPP (mean = 2.4 kg, standard deviation = 1.9). Using a Beta error of 0.2 and an Alpha error of 0.01, the sample size required for each group is 50, and assuming a 20% of the loss to follow up (based on the pilot study), and a 30% additional to ensure representativeness of the sample and power, the sample size will be incremented to 78 participants in each group, total sample size of 156 participants.

Randomization: Eligible participants will be randomly assigned to hybridized LSI or only DPP with 1:1 allocation.

Implementation:

Diabetes Prevention Program: The DPP Group Lifestyle Balance (GLB) core curriculum content modified from the original DPP is available online, in both English and Spanish. Despite the intent of facilitating T2D care for the U.S. Hispanic population, the advantage of the Spanish language version, and the robust and general recommendations in which the DPP GLB program is based, this effort was not a true transculturalization process. Important differences among various ethnocultural co-populations and environments were not addressed. For example, in Venezuela, there are unique culinary customs: units of measure during food preparation, types of whole foods in their natural form, and recipes with foods that are not easily available. In addition, recommendations of physical activities must be feasible for a certain population based on religious customs, social norms, the built environment, climate and terrain, and socioeconomic constraints; even, there are food patterns and behaviors regionally different in the same country.

The tDNA process was implemented in the following steps to undertake the transcultural adaptation of the DPP content: 1) Identification target population: adult's population in Venezuela. 2) Identification of the topic or research/clinical question: One out three adults in Venezuela has prediabetes. Evidence-based solutions are required to reduce diabetes burden in Venezuela. 3) Team of experts in the source (DPP) and target population (Venezuelan culture): A group of Venezuelan experts composed by four diabetologists, one primary care physician, and two community members trained and certificate by this team to provide T2D prevention programs implemented the adaptive content of the DPP GLB program. 4) Identification and resolution of cultural nodes using a framework: The DPP content was organized with the Ecological Validity Model (EVM). Using an interactive process each discrepancy between the content and cultural or local costumes were identified and modified in base to the EVM framework (e.g. recipes were adapted to the current socio-economic moment of the country). Finally, T2D prevention curriculum content was culturally adapted to Venezuelan adults avoiding any incongruence with the original version. Healthy options, goal settings, and problem-solving were consistent attributes of the culturally adapted program. Details of this transcultural adaptation will be published soon. This content was used in the pilot study.

Low-Energy Liquid-Diet (LELD): LELD, structured food reintroduction, and then a weight-loss maintenance program have demonstrated being a feasible and acceptable strategy to lose and maintain weight during 12 months. A "home-made" milk- and fruit-juice-based diet (811 kcal/day, 64 g protein, 132 g carbohydrate, 6 g fat) will be recommended. Recipes and preparation techniques were transculturally adapted to the population using local available low-cost foods in Venezuela. A pilot study assessing acceptability, appropriateness, and feasibility of this LELD strategy in Venezuelan adults with obesity is ongoing.

ELIGIBILITY:
Inclusion Criteria:

* Adults between 20 to 79 years years old
* No personal history of type 2 diabetes
* Body mass index ≥ 25 kg/m2
* High risk for type 2 diabetes

Exclusion Criteria:

* Chronic ischemic heart disease: acute myocardial infarction, stable angina, unstable angina.
* Stroke.
* Use of anticoagulants
* Severe renal failure
* Heart failure.
* Cannot do moderate-intensity physical activity
* Cannot attend most sessions
* Pregnancy or plans of having during the next sixth months
* Cancer or chemotherapy.
* Use of medications that affect weight (e.g. levothyroxine, pregabalin, orlistat)

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2021-11-23 (Actual); Study Completion 2022-01-15 (Actual)

PRIMARY OUTCOMES:
Change of weight in kilograms | 6 months
  The difference of change of weight in kilograms between the arms of the intervention

SECONDARY OUTCOMES:
Change in the points of Acceptance of the program assessed by a questionnaire using a Likert scale | 6 months
  The level of acceptance of the program will be measured with a questionnaire. Each question will be scored using a Likert scale from 0 to 5 points, where 0 is the worse and 5 is the best result. The change in the points of each question will be compared between arms of intervention.
Change in the points of Appropriateness of the core-curriculum assessed by a questionnaire using a Likert scale | 6 months
  The level of appropriateness of the core-curriculum will be measured with a questionnaire. Each question will be scored using a Likert scale from 0 to 5 points, where 0 is the worse and 5 is the best result. The change in the points of each question will be compared between arms of intervention.
Percentage of Attendance to the program | 6 months
  The percentage of attendance to the program will be calculated as the number of sessions that the participant attended from the total number of sessions. The percentage will be compared between arms of the intervention.
Percentage of Completion of the program. | 6 months
  The completion percentage will be measured as the percentage of participants that finalized the program. The percentage will be compared between arms of intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Juan P Gonzalez-R, MD, Principal Investigator — Foundation for Public Health and Epidemiological Research of Venezuela
Locations (2):
- Venezuela (2):
  - Maria M. Infante Garcia, Caracas, Chacao
  - FISPEVEN, Caracas, Chacao

IPD SHARING:
Plan to Share IPD: No
There is no plan to share data with other researchers

DOCUMENTS (1):
  • Study Protocol (2020-02-17): https://cdn.clinicaltrials.gov/large-docs/71/NCT04927871/Prot_000.pdf